CLINICAL TRIAL: NCT01435798
Title: Clinical Neuropharmacology of Pain in Spinal Cord Injury- Dextromethorphan Dose Response Clinical Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Christine N. Sang, MD, MPH, Director, Translational Pain Research, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2000p001387-A; R01NS041503 (NIH)
Record Dates: First submitted 2011-09-15; First posted 2011-09-19 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Central Neuropathic Pain; Allodynia; Spinal Cord Injury
Keywords: chronic pain; central neuropathic pain; spinal cord injury; dextromethorphan; lidocaine; combination therapy; analgesia
MeSH Terms: conditions — Hyperalgesia; Spinal Cord Injuries; Chronic Pain; Agnosia | interventions — Dextromethorphan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 0% MTD Dex (Placebo Comparator): 0% MTD Dextromethorphan
  Interventions: Drug: Dextromethorphan
- 25% MTD Dex (Experimental): 25% MTD Dextromethorphan
  Interventions: Drug: Dextromethorphan
- 50% MTD Dex (Experimental): 50% MTD Dextromethorphan
  Interventions: Drug: Dextromethorphan
- 100% MTD Dex (Experimental): 100% MTD Dextromethorphan
  Interventions: Drug: Dextromethorphan

INTERVENTIONS:
Drug: Dextromethorphan — 0, 25, 50 and 100% of maximum tolerated dose, each administered over a 4 week period

SUMMARY:
This randomized, placebo-controlled, double-blind 4x4 crossover clinical trial was part of a larger NIH-funded study to evaluate the analgesic efficacy of three doses of chronic oral (PO) dextromethorphan compared to placebo in central neuropathic pain following spinal cord injury. Subjects' maximally tolerated doses (MTD) were first determined to establish individual dose-analgesic response relationships in a run-in period; following a washout period, subjects were then randomized to receive an order of four doses of dextromethorphan (including placebo) in a 4x4 Latin square cross-over design.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female adults, age 18 to 70 with central neuropathic pain for a minimum of 3 months following SCI as confirmed by neurologic evaluation, with an average pain intensity score of at least moderate over at least 50% of the day for the 7 days prior to the screening visit and over the 7 days prior to starting study medication.
2. Subjects used no medication or a stabilized medication regimen for chronic and well-controlled medical conditions
3. Serum laboratory examination obtained at study entry:

   * Liver function tests (albumin within 20% of normal, SGOT/SGPT within 50% of normal).
   * For women of childbearing age: negative serum beta HCG.
4. Postmenopausal women, or be physically incapable of childbearing, or be practicing an acceptable method of birth control.
5. Normal cognitive function.
6. Normal communicative ability (English).
7. Ability to demonstrate competence in recording five times daily in pain diary for 1 week (with 100% compliance), and in completing required questionnaires.
8. Signed informed consent.

Exclusion Criteria:

1. Pregnancy or breast-feeding.
2. Renal or hepatic dysfunction.
3. Significant cardiac disease (e.g. MI within 1 year).
4. Signs or symptoms of central neurological disorder, excluding SCI.
5. Severe psychological disorder requiring treatment.
6. Concurrent use of monoamine oxidase inhibitors within 2 weeks prior to study entry.
7. Use of known CYP2D6 (but not CYP3A4) inhibitors or inducers.
8. History of hypersensitivity or intolerance to dextromethorphan or lidocaine.
9. Chronic substance abuse, including alcohol.
10. Participation in a study of an investigational drug or device within 30 days prior to screening for this study.
11. Poor metabolizer of P450 2D6 substrates.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2003-04; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine N. Sang, MD, MPH, Principal Investigator — Translational Pain Research, Brigham and Women's Hospital (Disclosure: Patent)
Locations (1):
- Translational Pain Research, Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- See also: Translational Pain Research, Brigham and Women's Hospital — http://www.paintrials.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited nationally from referring physicians, through advertisements, and through existing databases.
Pre-assignment Details: During the screening visit, P450 2D6 phenotype status was determined for each subject to identify drug-metabolizing capacity; those who were P450 2D6 poor-metabolizers were excluded. Following screen, each subject entered a dose escalation period to determine his/her maximum tolerated dose (MTD), prior to randomization.
Groups:
- Dextromethorphan Dose Response (DDR) Clinical Trial: Each subject received four doses of dextromethorphan; 0% (placebo), 25%, 50%, and 100% of the maximum tolerated dose in a balanced randomized order. Each dose was administered for a period of 28 days; on day 21 of each phase, subjects traveled to the study site to undergo study procedures in a nested clinical trial (not described here).
Period: Overall Study
Arm/Group | Dextromethorphan Dose Response (DDR) Clinical Trial
Started | 26 (Crossover design)
0% MTD | 25
25% MTD | 26
50% MTD | 25
100% MTD | 25
Completed | 25 (Crossover design)
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Dextromethorphan Dose Response Clinical Trial: Each subject received four doses of dextromethorphan; 0% (placebo), 25%, 50%, and 100% of the maximum tolerated dose in a balanced randomized order. Each dose was administered for a period of 28 days; on day 21 of each phase, subjects traveled to the study site to undergo study procedures in a nested clinical trial (not described here).
Arm/Group | Dextromethorphan Dose Response Clinical Trial
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.84 (11.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 12
Region of Enrollment [Number; unit: participants]
  North America | 26

OUTCOME MEASURES:

1. Primary Outcome: Mean Pain Intensity (Percent Change From Baseline)
Description: Primary outcome was percent change from baseline in mean pain intensity (transformed Gracely Scale; 0-35). Baseline was defined as the week prior to randomization. The greater the percent change, the bigger the reduction in pain intensity.
Time Frame: 1st week of maintenance period (week prior to hospital admission for nested study; subjects traveled to Boston on days 6-7 of the maintenance period)
Measure: Mean (Standard Error); unit: Percent change from baseline
Groups:
- 0% MTD Dex: 0% (placebo) of maximum tolerated dose of dextromethorphan; dose was administered for a period of 28 days, and on day 21, subjects traveled to the study site to undergo additional study procedures.
- 25% MTD Dex: 25% of maximum tolerated dose of dextromethorphan; dose was administered for a period of 28 days, and on day 21, subjects traveled to the study site to undergo additional study procedures.
- 50% MTD Dex: 50% of maximum tolerated dose of dextromethorphan; dose was administered for a period of 28 days, and on day 21, subjects traveled to the study site to undergo additional study procedures.
- 100% MTD Dex: 100% of maximum tolerated dose of dextromethorphan; dose was administered for a period of 28 days, and on day 21, subjects traveled to the study site to undergo additional study procedures.
Arm/Group | 0% MTD Dex | 25% MTD Dex | 50% MTD Dex | 100% MTD Dex
Number analyzed (Participants) | 25 | 26 | 25 | 25
Percent change from baseline | -0.006 (0.01) | -0.018 (0.005) | -0.073 (0.01) | -0.24 (0.01)

2. Secondary Outcome: Satisfaction
Description: Satisfaction with study treatment assessed over the 7 days prior to admission (5-point categorical scale)
Time Frame: Last week prior to admission (end of 1-week maintenance period)
Measure: Count of Participants; unit: Participants
Arm/Group | 0% MTD Dex | 25% MTD Dex | 50% MTD Dex | 100% MTD Dex
Number analyzed (Participants) | 25 | 26 | 25 | 25
Participants
  Not Satisfied | 20 | 18 | 16 | 9
  Fairly Satisfied | 2 | 5 | 7 | 8
  Satisfied | 3 | 2 | 0 | 5
  Very/Extremely Satisfied | 0 | 1 | 2 | 3

ADVERSE EVENTS:
Time Frame: Adverse event data were collected post-dose through the end of treatment in each arm.
Description: All anticipated and unanticipated post-dose adverse events that were possibly, probably, or definitely related to the study drug are reported.
Arm/Group | 0% MTD Dex | 25% MTD Dex | 50% MTD Dex | 100% MTD Dex
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/26 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 2/25 | 3/26 | 2/25 | 16/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0% MTD Dex (N=25) | 25% MTD Dex (N=26) | 50% MTD Dex (N=25) | 100% MTD Dex (N=25)
Tinnitis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) — Not present at baseline, defined as:1) prior to randomization, in DDR; 2) Prior to lido infusion, on 100% Dex, in D/L. In DDR, all AEs were of mild intensity. In D/L, AEs were assessed at Cmax and were >= mild. No infusions were terminated for AEs.
Sedation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 8 (8) — Not present at baseline, defined as:1) prior to randomization, in DDR; 2) Prior to lido infusion, on 100% Dex, in D/L. In DDR, all AEs were of mild intensity. In D/L, AEs were assessed at Cmax and were >= mild. No infusions were terminated for AEs.
Blurry Vision (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Interference with Alertness (Nervous system disorders) | 2 (2) | 3 (3) | 0 (0) | 3 (3)
Interference with Ability to Drive (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No